CLINICAL TRIAL: NCT03376503
Title: A Randomized, Double-blind, Parallel Study Comparing Pharmacokinetic (PK) and Pharmacodynamic (PD) Parameters of Pegcyte (Nanogen) and Reference Product Neulastim (Roche) for Chemotherapy-induced Neutropenia in Breast-cancer Patients
Brief Title: Nanogen Pegfilgrastim (Pegcyte) PK/PD Clinical Study in Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanogen Pharmaceutical Biotechnology Joint Stock Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NNG04
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pegcyte (Nanogen pegfilgrastim) (Experimental): pegcyte 6 mg in the first cycle
  Interventions: Drug: Pegfilgrastim
- Neulastim (Roche pegfilgrastim) (Active Comparator): Neulastim 6 mg in the first cycle
  Interventions: Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Pegfilgrastim — PK,PD and safety assessment

SUMMARY:
Breast cancer patients scheduled to receive myelosuppressive chemotherapy (AC regimen) will be enrolled in this study. Eligible patients receive single SC injection of pegcyte or neulastim 24 hours after administration of chemotherapy (Doxorubicin and Cyclophosphamide) in the first cycle (14 days each cycle). Blood samples are collected to determine the serum concentration of investigational drugs at specific time points in the first cycle. Absolute neutrophil count, CD34+ count, Cmax (maximum serum concentration), AUC0-t (area under the curve of the plasma concentration time) and Tmax (time required to reach Cmax) will be calculated from the serum concentration profile

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 - 65 years.
* Patients with histological confirmed primary invasive breast cancer; stage I, II or III.
* Patients had no prior chemotherapy treatments.
* Patients scheduled to undergo myelosuppressive Doxorubicin and Cyclophosphamide chemotherapy for 04 cycles, and Paclitaxel chemotherapy for the next 04 cycles; patients were available for 14 days of each cycle for the first 03 chemotherapy cycles.
* Patients with baseline ANC ≥ 1.5 x 109/L, PLT ≥ 100 x 109/L, HgB ≥ 9 g/dL, WBC ≥ 3,000/mL and albumin ≥ 3.0 g/dL.
* Performance status as per ECOG (Eastern Cooperative Oncology Group) score 0, 1 or 2.
* Willing to give written and signed informed consent

Exclusion Criteria:

* Patients with prior exposure of G-CSF or GM-CSF or its pegylated products in clinical development less than 6 months prior to randomization.
* Myelotoxic concomitant treatment such as chloramphenicol, methotrexate, immunomodulating agents, interferons during 10 days before randomization.
* Received systemic antibiotic treatment within 72 hours of chemotherapy.
* Chronic use of corticosteroids, prior bone marrow or stem cell transplant.
* Patients who had an immediate/ concurrent exposure to radiotherapy or surgery (within 4 weeks).
* Severe medical disease: cardiovascular, hepatic, renal, pulmonary…
* Known cases of hematological disease (sickle cell anemia, AML…)
* History of HIV positive, active hepatitis.
* Pregnant and lactating women or patients planning to become pregnant.
* Known allergic reactions to study medications.
* Positive to anti-pegfilgrastim antibody test.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 24 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time 0 to the last time point (AUC0-t) for serum Pegfilgrastim (PEG-GCSF) | day 2 (0h, 3h, 6h, 12±4h), day 3 (24h), day 4 (48h), day 5 (72h), day 7 (120h), day 8 (144h), day 9 (168h), day 11 (216h), and day 14 (288h) of the first cycle
  (AUC0-t)

SECONDARY OUTCOMES:
Apparent clearance (CL) for serum Pegfilgrastim | day 2 (0h, 3h, 6h, 12±4h), day 3 (24h), day 4 (48h), day 5 (72h), day 7 (120h), day 8 (144h), day 9 (168h), day 11 (216h), and day 14 (288h) of the first cycle
Maximum concentration (Cmax) for serum Pegfilgrastim | day 2 (0h, 3h, 6h, 12±4h), day 3 (24h), day 4 (48h), day 5 (72h), day 7 (120h), day 8 (144h), day 9 (168h), day 11 (216h), and day 14 (288h) of the first cycle
Half-life (T½) for serum Pegfilgrastim (PEG-GCSF) | day 2 (0h, 3h, 6h, 12±4h), day 3 (24h), day 4 (48h), day 5 (72h), day 7 (120h), day 8 (144h), day 9 (168h), day 11 (216h), and day 14 (288h) of the first cycle
Area under the serum concentration-time curve (AUC0-inf) of Pegfilgrastim | day 2 (0h, 3h, 6h, 12±4h), day 3 (24h), day 4 (48h), day 5 (72h), day 7 (120h), day 8 (144h), day 9 (168h), day 11 (216h), and day 14 (288h) of the first cycle
Time to maximum concentration (Tmax) for serum Pegfilgrastim | day 2 (0h, 3h, 6h, 12±4h), day 3 (24h), day 4 (48h), day 5 (72h), day 7 (120h), day 8 (144h), day 9 (168h), day 11 (216h), and day 14 (288h) of the first cycle
Terminal elimination rate constant (λz) for serum Pegfilgrastim | day 2 (0h, 3h, 6h, 12±4h), day 3 (24h), day 4 (48h), day 5 (72h), day 7 (120h), day 8 (144h), day 9 (168h), day 11 (216h), and day 14 (288h) of the first cycle
Maximum change in CD34+ count | day 2 (0h), day 5 (72h), day 7 (120h), and day 8 (144h) of the first cycle.
Area under the curve above baseline of ANC [ANC_AUC(0-tlast)] | day 2 (0h, 3h, 6h, 12±4h), day 3 (24h), day 4 (48h), day 5 (72h), day 7 (120h), day 8 (144h), day 9 (168h), day 11 (216h), and day 14 (288h) of the first cycle
Time of maximum change from baseline for ANC in days (ANC_Tmax) | day 2 (0h, 3h, 6h, 12±4h), day 3 (24h), day 4 (48h), day 5 (72h), day 7 (120h), day 8 (144h), day 9 (168h), day 11 (216h), and day 14 (288h) of the first cycle
Maximum change from baseline in absolute neutrophil count from time 0 to the last time point ANC AUC0-t | day 2 (0h, 3h, 6h, 12±4h), day 3 (24h), day 4 (48h), day 5 (72h), day 7 (120h), day 8 (144h), day 9 (168h), day 11 (216h), and day 14 (288h) of the first cycle
Maximum change from baseline in absolute neutrophil count (ANC); ANC_Cmax | day 2 (0h, 3h, 6h, 12±4h), day 3 (24h), day 4 (48h), day 5 (72h), day 7 (120h), day 8 (144h), day 9 (168h), day 11 (216h), and day 14 (288h) of the first cycle
Incidence of adverse events | cycle 1 from day 2 to day 14
  Including changes in vitals and laboratory investigations

CONTACTS AND LOCATIONS:
Locations (1):
- Vietnam National Cancer Institute (Hospital K), Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided